CLINICAL TRIAL: NCT04758364
Title: Factors That Effect the Gait Speed in Diabetic Individuals Without Neuropathy
Status: Completed | Type: Observational
Sponsor: GULIN FINDIKOGLU (Other)
Responsible Party: Sponsor-Investigator, GULIN FINDIKOGLU, Assoc Proffessor, MD, PhD, Pamukkale University
Organization: Pamukkale University (Other)
Other Study IDs: 60116787-020/75097
Record Dates: First submitted 2021-02-11; First posted 2021-02-17 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Gait Disorder, Sensorimotor; Diabetes Mellitus, Type 2
Keywords: Mini-Mental State Examination; gait; aerobic capacity; HbA1c; muscle; hypertension; glucose
MeSH Terms: conditions — Gait Disorders, Neurologic; Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: measurement of gait speed — Cross sectional, cohort
  Other Names: measurement of aerobic capacity; measurement of muscle mass; measurement of blood glucose and HbA1c; cognitive function testing; physical activity questioning; blood pressure measurement

SUMMARY:
This study planned to investigate the role of potential explanatory factors effecting the speed of gait such as muscle mass, aerobic capacity, physical activity status, cognitive function, blood pressure, and metabolic measures considering age, sex, and education years in diabetic individuals without neuropathy.

DETAILED DESCRIPTION:
Type 2 diabetic people will be screened by clinical symptoms of neuropathy and DN4 questionnaire. Among those who did not have neuropathic symptoms or who have DN4 score below 4 will be considered for the study.Then aerobic capacity will be measured by a cycle ergometer and VO2max will be obtained. Weight, body mass index and muscle mass will be measured by bioimpedance analysis. Physical activity status will be determined by International Physical Activity Score (IPAQ). Cognitive function will be evaluated by Mini Mental test. HbA1c and fasting blood glucose will be measured in venous blood after overnight fasting. Blood pressure will be measured in the sitting position after resting from the left arm. Speed of gait will be measured by an accelerometer.Then, the effect of above mentioned factors on speed of gait will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with Diabetes Mellitus less than 10 years but longer than 1 year
* Absence of neuropathic symptoms
* DN4 questionnaire sore less than 4

Exclusion Criteria:

Individuals who had

* insulin therapy,
* poor glycemic control,
* manifesting cardiovascular disease,
* retinopathy or other visual problems,
* diabetic neuropathy,
* nephropathy,
* cerebrovascular disease,
* cognitive impairment,
* heart failure,
* alcohol or cigarette dependence,
* cancer,
* chemo/radiotherapy,
* foot ulcer,
* orthopedical or surgical problems
* wheel-chair or any assistive devices for ambulation
* prominent knee or hip arthritis, prosthesis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 Diabetic individuals without neuropathy
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
gait speed | The gait speed will be measured once within a month after the participants enrolled.
  gait speed measured by wearable accelerometer

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No